CLINICAL TRIAL: NCT07276685
Title: Evaluation of the Success of TheraCal PT and Biodentine in Pulpotomy Treatment of Primary Teeth and the Effect of Low-Level Laser Therapy (LLLT) on Treatment Outcomes
Brief Title: Evaluation of the Success of TheraCal PT in Pulpotomy Treatment of Primary Teeth Using Low-Level Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NECIBE DAMLA ŞAHIN (Other)
Collaborators: Tokat Gaziosmanpasa University (Other)
Responsible Party: Sponsor-Investigator, NECIBE DAMLA ŞAHIN, Assistant Professor, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/92; 2022/92 (Other: Tokat Gaziosmanpasa University, BAP Unit)
Record Dates: First submitted 2025-11-18; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Primary Tooth Pulpotomy; Vital Pulp Therapy
Keywords: Primary Tooth; Pulpotomy; TheraCal PT; Biodentine; Low-Level Laser Therapy
MeSH Terms: interventions — Biocompatible Materials; Low-Level Light Therapy; Lasers

STUDY DESIGN:
Intervention Model Description: The study was designed as a parallel-group randomized clinical trial. Sixty primary molars from children aged 4-9 years were randomly assigned to four intervention groups according to the material used (Biodentine or TheraCal PT) and the use of low-level laser therapy (LLLT).
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded to the treatment groups during clinical and radiographic evaluations. Participants and operators were not blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Biodentine (Active Comparator): Primary molars treated with pulpotomy using Biodentine without low-level laser therapy (LLLT). After coronal pulp removal, Biodentine (Septodont, France) was placed over the remaining pulp tissue. No laser application was performed.
  Interventions: Procedure: Biodentine Pulpotomy
- LLLT + Biodentine (Experimental): Primary molars treated with Biodentine pulpotomy combined with low-level laser therapy. After pulpotomy, diode laser (940 nm, 10 s, non-contact mode) was applied over the pulp chamber floor, followed by placement of Biodentine (Septodont, France).
  Interventions: Device: Low-Level Laser Therapy + Biodentine
- TheraCal PT (Experimental): Primary molars treated with pulpotomy using TheraCal PT without low-level laser therapy. After coronal pulp removal, TheraCal PT (Bisco Inc., USA) was applied directly onto the pulp tissue. No laser application was performed.
  Interventions: Procedure: TheraCal PT Pulpotomy
- LLLT + TheraCal PT (Experimental): Primary molars treated with TheraCal PT pulpotomy combined with low-level laser therapy. Following pulpotomy, a 940 nm diode laser (Biolase, USA) was applied for 10 seconds in non-contact mode, followed by application of TheraCal PT (Bisco Inc., USA).
  Interventions: Device: Low-Level Laser Therapy + TheraCal PT

INTERVENTIONS:
Procedure: Biodentine Pulpotomy — After coronal pulp removal, Biodentine (Septodont, France) was placed over the remaining pulp tissue. No laser application was performed.
  Other Names: biomaterial
  Arms: Biodentine
Device: Low-Level Laser Therapy + Biodentine — After pulpotomy, diode laser (940 nm, 10 s, non-contact mode) was applied over the pulp chamber floor, followed by placement of Biodentine (Septodont, France).
  Other Names: Laser and biomaterial
  Arms: LLLT + Biodentine
Procedure: TheraCal PT Pulpotomy — After coronal pulp removal, TheraCal PT (Bisco Inc., USA) was applied directly onto the pulp tissue. No laser application was performed.
  Arms: TheraCal PT
Device: Low-Level Laser Therapy + TheraCal PT — Following pulpotomy, a 940 nm diode laser (Biolase, USA) was applied for 10 seconds in non-contact mode, followed by application of TheraCal PT (Bisco Inc., USA).
  Arms: LLLT + TheraCal PT

SUMMARY:
This randomized clinical study aimed to compare the clinical and radiographic outcomes of TheraCal PT and Biodentine in pulpotomy treatment of primary teeth and to evaluate the influence of low-level laser therapy (LLLT) on treatment outcomes in pediatric patients.

DETAILED DESCRIPTION:
This prospective randomized clinical trial was conducted at Tokat Gaziosmanpaşa University, Faculty of Dentistry, Department of Pediatric Dentistry. The study included healthy children aged 4 to 9 years who required pulpotomy treatment for primary molar teeth.

Eligible teeth were randomly allocated into four groups according to the pulpotomy material used and the application of low-level laser therapy (LLLT): (1) Biodentine, (2) LLLT + Biodentine, (3) TheraCal PT, and (4) LLLT + TheraCal PT.

Low-level laser therapy was performed using a 940 nm diode laser in non-contact mode immediately after coronal pulp removal. All treated teeth were restored with stainless steel crowns. Clinical and radiographic evaluations were scheduled at baseline and at 3, 6, and 12 months follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

Healthy children aged between 6 and 9 years. Primary molars with carious exposures requiring pulpotomy treatment. Teeth with vital pulp confirmed by the absence of spontaneous pain and the presence of normal bleeding after coronal pulp removal.

Teeth with restorable crowns suitable for stainless steel crown restoration. Cooperative patients who can attend all follow-up appointments.

Exclusion Criteria:

Teeth with signs of irreversible pulpitis or necrosis (e.g., spontaneous or nocturnal pain).

Teeth with internal or external root resorption, furcal or periapical radiolucency.

Non-restorable teeth or those with excessive loss of crown structure. Patients with systemic diseases or on long-term medication that could affect healing.

Uncooperative children or those lost to follow-up.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Clinical and Radiographic Success Rate of Pulpotomy Treatments in Primary Molars | 12 months after treatment
  Number of teeth with clinical success defined as absence of spontaneous pain, swelling, sinus tract, pathological mobility, or tenderness to percussion, and number of teeth with radiographic success defined as absence of internal or external root resorption and absence of furcal or periapical radiolucency. Results will be reported as number and percentage of successful teeth.

SECONDARY OUTCOMES:
Interim Clinical and Radiographic Success Rates | 3 and 6 months after treatment
  Number of teeth meeting clinical and radiographic success criteria at interim follow-up visits, reported as number and percentage of successful teeth.
Effect of Low-Level Laser Therapy (LLLT) on Pulpotomy Success | 12 months after treatment
  Difference in the proportion of clinically and radiographically successful teeth between the laser-treated groups and non-laser groups, expressed as number and percentage of successful teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Necibe Damla ŞAHİN, DDS, PhD, Principal Investigator — Tokat Gaziosmanpaşa University, Faculty of Dentistry, Department of Pediatric Dentistry, Tokat, Turkey
Locations (1):
- Tokat Gaziosmanpasa University Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study involved pediatric participants and the data contain potentially identifiable information. Only summary data will be available in the published article.